CLINICAL TRIAL: NCT06182761
Title: Efficacy and Safety of Sunvozertinib With Anlotinib in EGFR-TKIs Resistant EGFR-sensitive Mutated Locally Advanced or Metastatic Non-small Cell Lung Cancer (NSCLC): a Prospective, Single-arm, Phase II Trial
Brief Title: A Study of Sunvozertinib Combined With Anlotinib in Local Advanced or Metastatic Non-small Cell Lung Cancer
Acronym: WUKONG-9
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Shanghai Zhongshan Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: WUKONG9
Record Dates: First submitted 2023-12-01; First posted 2023-12-27 (Actual); Last update posted 2023-12-27 (Actual); Status verified 2023-12

CONDITIONS: NSCLC
MeSH Terms: interventions — anlotinib

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- sunvozertinib in combination with Anlotinib (Experimental)
  Interventions: Drug: Sunvozertinib combination with Anlotinib

INTERVENTIONS:
Drug: Sunvozertinib combination with Anlotinib — Sunvozertinib 300 mg once daily (QD) with Anlotinib 12mg once daily （QD in Day 1-14） ，21 days in one cycle.

SUMMARY:
The study will evaluate the efficacy and safety of treatment with sunvozertinib in combination with Anlotinib in patients whose disease has progressed following first-line EGFR-TKIs treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Capable of giving signed informed consent, which includes compliance with the requirements and restrictions listed in the informed consent form and in this protocol.
2. Pathologically confirmed non-squamous NSCLC. Locally advanced or metastatic NSCLC
3. EGFR sensitive mutations confirmed by accredited local laboratories， including 19del、L858R and T790M。
4. Intolerant or refuses, or not suitable for systemic chemotherapy.
5. Progressed after EGFR-TKI targeted therapy or are intolerant to standard treatment; if carry T790M mutation, need to be treated with osimertinib or other third-generation EGFR-TKI.
6. World Health Organization performance status of 0 to 1
7. Life expectancy >12 weeks at Day 1.
8. At least 1 lesion to be measured
9. Females must be using highly effective contraceptive measures, and must have a negative pregnancy test prior to start of dosing if of childbearing potential, or must have evidence of non-childbearing potential by fulfilling criteria at screening.
10. Male patients must be willing to use barrier contraception

Exclusion Criteria:

1. Any known RET rearrangement, BRAF V600E mutation, NTRK fusion, MET ex14 skip mutation, MET amplification (defined as tissue detection GCN ≥ 5 by NGS)
2. Any concurrent and/or other active malignancy within 2 years
3. Major surgery within 4 weeks of the first dose of IP
4. Any unresolved toxicities from prior therapy.
5. Past medical history of ILD (interstitial lung disease)/pneumonitis, drug-induced ILD/pneumonitis, radiation pneumonitis that required steroid treatment, or any evidence of clinically active ILD/pneumonitis
6. Any evidence of severe or uncontrolled systemic diseases.
7. Any of the following cardiac criteria:

   i) Mean resting QTc >470 msec ii) Any clinically important abnormalities in rhythm, conduction, or morphology of resting electrocardiogram iii) Any factors that increase the risk of QTc prolongation or risk of arrhythmic events
8. Refractory nausea and vomiting, chronic gastrointestinal diseases, inability to swallow the formulated product, or previous significant bowel resection that would preclude adequate absorption of Sunvozertinib and Anlotinib
9. Severe allergies to Sunvozertinib and Anlotinib

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2024-01 (Estimated); Primary Completion 2026-01 (Estimated); Study Completion 2028-07 (Estimated)

PRIMARY OUTCOMES:
ORR | initiate from first dose until the date of confirmed response, assessed up to 24 weeks
  Objective response rate (ORR) as assessed by the investigator according to RECIST 1.1 criteria.

SECONDARY OUTCOMES:
PFS | initiate from first dose, every 6 weeks until PD or study close, an average of 1 year
  PFS as assessed by the investigator according to RECIST 1.1
OS | through study completion, an average of 1.5 years
  initiate from first dose to death from any cause
DoR | an average of 1 year
  The period from the first judgment of CR or PR to PD
AE | through study completion, an average of 1 year
  TRAE as assessed by the investigator according to CTCAE 5.0